CLINICAL TRIAL: NCT05466032
Title: Exploring the Evolution of the Mind-body Connection as First-year Osteopathic Medical Students Learn About Common Osteopathic Dysfunctions
Brief Title: Evolution of the Mind-body Connection While Learning About Common Osteopathic Dysfunctions
Status: Completed | Type: Observational
Sponsor: Mikhail Volokitin, MD, DO. (Other)
Responsible Party: Sponsor-Investigator, Mikhail Volokitin, MD, DO., Associate Professor OMM Department Touro College, The Touro College and University System
Organization: The Touro College and University System (Other)
Other Study IDs: TouroCOM-OMM
Record Dates: First submitted 2022-07-16; First posted 2022-07-20 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Medical School Syndrome; Mind Body Awareness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First year TouroCOM osteopathic medical students: As required by the Touro College of Osteopathic Medicine curriculum, all first year osteopathic students are enrolled in Osteopathic Manual Manipulation (OMM). This course meets three hours per week for the duration of the school year and teaches students about different osteopathic dysfunctions, as well as techniques for how to treat them.
  Interventions: Other: Osteopathic Manual Manipulation (OMM) Curriculum
- Master of Science TouroCOM students: Students enrolled in the Master of Science in Interdisciplinary Studies in Biological and Physical Sciences at TouroCOM complete almost all of the same courses as the osteopathic medical students, but are not exposed Osteopathic Manual Manipulation (OMM). This cohort will act as the control as they undergo similar environmental stress, but will not learn about common osteopathic dysfunctions or their treatments.

INTERVENTIONS:
Other: Osteopathic Manual Manipulation (OMM) Curriculum — Osteopathic medical students are enrolled in the OMM curriculum while masters students are not enrolled.
  Groups: First year TouroCOM osteopathic medical students

SUMMARY:
Anecdotally, as first-year medical students learn about common osteopathic dysfunctions, they seem to become more aware of possible dysfunctions in their own bodies. This study will explore whether this new awareness is because of a strengthened mind-body connection, leading to increased proprioceptive awareness, or whether these students are experiencing "medical student syndrome." Medical school syndrome is a common phenomenon, especially in the first years of medical school, defined as experiencing "vague bodily symptoms in terms of the latest disease they have learnt about."

This study will be conducted in multiple phases throughout 2022- 2023, based around the first year Osteopathic Manual Manipulation (OMM) exam schedule. After study recruitment during orientation week, first year students will be given the baseline participant survey. This survey asks participants to report pain/discomfort in the thoracic, lumbar, or rib/chest areas, as well as what this sensation may be attributed to (ex: somatic dysfunction, muscle soreness, traumatic injury, etc.). After completing the surveys, participants will undergo an osteopathic evaluation to confirm their stated symptoms. Researchers will not be aware of the participants' survey answers for the duration of the data collection portion of the study to reduce unintentional bias during the osteopathic evaluations.

After the first-year students complete each OMM module (thoracic spine, lumbar spine, ribs/chest), they will be given the same survey and osteopathic evaluation. Timing is of particular importance in this study-- conducting the survey and evaluation at a time when students are acutely aware of somatic dysfunctions specific to each region will allow us to link acquisition of this knowledge to the mind-body connection. If a participant reports new or increased pain/discomfort in the region just taught, it is likely to be linked to an increased awareness of the region. The osteopathic evaluation, in conjunction with the participant's attribution of the sensation, will determine if the student is experiencing increased proprioception, or a case of medical school syndrome.

DETAILED DESCRIPTION:
Data collection will take place in three week-long phases over the course of the first semester, timed around each first year Osteopathic Manual Manipulation Course exam. In the week after the first-year exam, participants will undergo an osteopathic examination and fill out a questionnaire. This process should take approximately 30 minutes per session, for a total of 1.5 hours over the course of five months.

Data analysis will be conducted in the second semester. In total, the estimated period of time for this project will be from the last week in July 2022 to May 2023. This data analysis will involve matching student surveys given throughout the year with findings from the osteopathic evaluations. Comparing the baseline and the subsequent subject surveys during data analysis will allow researchers to identify whether a new somatic dysfunction has arisen during the research period, and whether the subject is able to correctly identify and attribute this dysfunction.

All participants will be coded both on the participant survey and the osteopathic evaluation data form to protect their anonymity, as well as to blind the researchers. Data will be stored in a Google Drive via Google Forms. Only the researchers will have access to these files via their Touro emails. There will not be any risk to participants, nor will there likely be much benefit to the participants after completing the study besides assisting in furthering the field of osteopathic research.

ELIGIBILITY:
Inclusion Criteria:

* student at TouroCOM Harlem

Exclusion Criteria:

* any current and significant musculoskeletal disorders, either chronic or acute
* pregnant or plans to become pregnant within the next six months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: First year osteopathic students enrolled at Touro College of Osteopathic Medicine Harlem as well as students enrolled in Touro's Master of Science Program in Interdisciplinary Studies in Biological and Physical Sciences
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2025-04-12 (Actual); Study Completion 2025-04-12 (Actual)

PRIMARY OUTCOMES:
Difference in Mind Body Connection | Assessed three times over the course of the semester after the initial baseline evaluation. Each assessment will be scheduled around the relevant first year Osteopathic Manual Manipulation exams.
  A change in proprioceptive abilities of first year medical students after learning about Osteopathic Manual Manipulation (OMM). This connection will be measured by comparing the participant's stated symptoms on a participant survey to the participant's stated attribution of the pain. If the pain is attributed correctly to a common somatic dysfunction recently learned by the student, as confirmed by an osteopathic evaluation performed by the researchers, then it will show an increase in bodily awareness that correlates with an accumulation of osteopathic knowledge.
Changed Incidence of Medical School Syndrome | Assessed three times over the course of the semester after the initial baseline evaluation. Each assessment will be scheduled around the relevant first year Osteopathic Manual Manipulation exams.
  A change in reported "vague bodily symptoms in terms of the latest disease they [students] have learnt about." The incidence of medical school syndrome will be assessed by comparing the participant survey to the findings of the osteopathic evaluation. If no dysfunctions are found during the evaluation, but are 1) reported on the participant survey and 2) attributed to a common, or uncommon, somatic dysfunction that had been taught in the first year TouroCOM OMM curriculum, it is a case of medical school syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Volokitin, MD, DO, Principal Investigator — Touro College of Osteopathic Medicine
Locations (1):
- Touro College of Osteopathic Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No specific individual participant data will be shared, only study tools (consent form, surveys, data collection tools) without participant information will be shared upon request.

REFERENCES:
- [Background] Woods SM, Natterson J, Silverman J. Medical students' disease: hypochondriasis in medical education. J Med Educ. 1966 Aug;41(8):785-90. No abstract available. PMID 4380602
- [Background] Lesho EP. An overview of osteopathic medicine. Arch Fam Med. 1999 Nov-Dec;8(6):477-84. doi: 10.1001/archfami.8.6.477. PMID 10575385
- [Background] Licciardone JC, Schultz MJ, Amen B. Osteopathic Manipulation in the Management of Chronic Pain: Current Perspectives. J Pain Res. 2020 Jul 20;13:1839-1847. doi: 10.2147/JPR.S183170. eCollection 2020. PMID 32765058
- [Background] Kuchera ML. Osteopathic manipulative medicine considerations in patients with chronic pain. J Am Osteopath Assoc. 2005 Sep;105(9 Suppl 4):S29-36. PMID 16249364
- [Background] Ezmeirlly HA, Farahat FM. Illness anxiety disorder and perception of disease and distress among medical students in western Saudi Arabia. Saudi Med J. 2019 Nov;40(11):1144-1149. doi: 10.15537/smj.2019.11.24654. PMID 31707412
- [Background] Moss-Morris R, Petrie KJ. Redefining medical students' disease to reduce morbidity. Med Educ. 2001 Aug;35(8):724-8. doi: 10.1046/j.1365-2923.2001.00958.x. PMID 11489098
- [Background] Salkovskis PM, Rimes KA, Warwick HM, Clark DM. The Health Anxiety Inventory: development and validation of scales for the measurement of health anxiety and hypochondriasis. Psychol Med. 2002 Jul;32(5):843-53. doi: 10.1017/s0033291702005822. PMID 12171378
- [Background] Szczurek K, Furgal N, Szczepanek D, Zaman R, Krysta K, Krzystanek M. "Medical Student Syndrome"-A Myth or a Real Disease Entity? Cross-Sectional Study of Medical Students of the Medical University of Silesia in Katowice, Poland. Int J Environ Res Public Health. 2021 Sep 19;18(18):9884. doi: 10.3390/ijerph18189884. PMID 34574807